CLINICAL TRIAL: NCT02642146
Title: Treatment of Digital Ulcers in Korean Patients With Systemic Sclerosis: a Prospective Cohort Study
Status: Terminated | Type: Observational
Why Stopped: We decided to terminate recruit earlier because patient recruiting was not active as expected at the beginning of the study.
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Eun Bong Lee, Professor/M.D, PhD, Seoul National University Hospital
Other Study IDs: SNUH-IMJ-002
Record Dates: First submitted 2015-12-24; First posted 2015-12-30 (Estimated); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Raynaud Disease; Systemic Sclerosis; Digital Ulcer
MeSH Terms: conditions — Raynaud Disease; Scleroderma, Systemic; digital ulcers | interventions — Calcium Channel Blockers; Phosphodiesterase Inhibitors; Prostaglandins

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years

INTERVENTIONS:
Drug: Calcium Channel Blockers
Drug: Phosphodiesterase Inhibitors
Drug: Endothelin receptor blocker
Drug: Prostanoids
Drug: Other vasodilator

SUMMARY:
This study evaluates the efficacy and safety of routine medical treatments of digital ulcers in patients with systemic sclerosis in a prospective cohort study.

DETAILED DESCRIPTION:
Systemic sclerosis (SSc) is a chronic autoimmune disease of unknown etiology with high morbidity and mortality. SSc manifests by fibrosis of skin and internal organs. Although the underlying mechanisms are still subject to investigation, endothelial dysfunction and abnormal immune response are thought to contribute to vascular dysfunction and fibrosis in SSc.

A hallmark feature of SSc is the presence of Raynaud phenomenon (RP) that is caused by reversible vasoconstriction of digital arteries triggered by exposure to cold or emotional stress. In up to 33-43% of SSc patients, the ischemia can progress to digital ulcers (DUs), which are often associated not only with pain but also with severe limitation in the daily activity, anxiety and depression among others. In severe cases, RP can be complicated by superinfection or gangrene, requiring surgical amputation.

The mainstay treatment of RP is restoration of the decreased blood flow using calcium channel blocker, protstanoids, phosphodiesterse V inhibitor, and endothelin receptor blocker. However, the efficacy and safety of those medications in RP-associated ulcers have not been definitive, especially in Korean patients with SSc. In addition, it remains unknown whether Korean SSc patients respond better to a treatment over others.

Study aims include

1. To establish a new prospective cohort of SSc patients with DU in Korea..
2. To investigate the current situation of SSc patients in Korea.
3. To investigate and compare the efficacy and safety of current medical treatments of DU in SSc patients in Korea

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 years or older
* SSc diagnosis according to 1980 or 2013 ACR classification criteria
* 1 or more active DU
* Patients who start or change medical treatment for DU
* Patients who are willing to participate

Exclusion Criteria:

* Pregnancy or active breast feeding
* Patients with life expectancy < 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with systemic sclerosis
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Time to resolution of cardinal DU | weeks or days (from baseline)

SECONDARY OUTCOMES:
Change in size of cardinal DU from baseline | weeks 4, 8, 12, 24 weeks
Change in DU number from baseline | weeks 4, 8, 12, 24
Number of new DU | weeks 4, 8, 12, 24
Case of successful digital ulcer treatment with tolerable side | weeks 4, 8, 12, 24
Number of patients with superinfection | weeks 4, 8, 12, 24

OTHER OUTCOMES:
Number of patients requiring amputation | weeks 4, 8, 12, 24
Number of adverse events | weeks 4, 8, 12, 24

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea